CLINICAL TRIAL: NCT04727411
Title: In Vivo Imaging and Impression Cytology Analysis of Conjunctival Changes as Potential Indicators for Ab-interno Gelatin Microstent Implantation Surgery Outcomes
Brief Title: Analysis of Conjunctival Changes as Indicators for Ab-interno Gelatin Microstent Implantation Surgery Outcomes
Acronym: IIT_XEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Néstor Ventura, Investigator, Glaucoma Department, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HCB/2019/0035
Record Dates: First submitted 2021-01-16; First posted 2021-01-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Glaucoma; Glaucoma Open-Angle Primary
Keywords: Gel stent; Trabeculectomy; In vivo confocal microscopy; Conjunctival impression cytology; Anterior segment optical coherence tomography
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gel Stent implantation (Experimental): XEN gel stent: a clear cornea incision in the inferotemporal quadrant was performed, injecting the XEN 45 device into the superonasal quadrant using an ab interno approach. Approximately 15 min before inserting the implant, 0.1 ml of a MMC solution (0.01%) was injected into the superior conjunctiva. Both stand-alone and combined phaco-glaucoma procedures were used.
  Interventions: Procedure: XEN45 Gel stent
- Trabeculectomy (Experimental): Trabeculectomy: the surgical technique is as follows: retro/peribulbar o subtenon's anesthesia, superior corneal traction suture, phacoemulsification through 2.2 with in-the-bag IOL implantation, a fornix-based conjunctival flap, sufficient but not excessive cauterization, application MMC 0,2 mg/ml for 2 minutes under the conjunctiva, then MMC was washed out with 100 ml of saline solution, then a scleral flap (4x3 mm in the trabeculectomy) is dissected. A sclerectomy with punch and peripheral iridectomy were performed, and suture nylon 10/00 sutures was used to place 3 or 4 stiches in the scleral flap
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: XEN45 Gel stent — XEN Gel stent implantation either combined or as a stand-alone procedure
  Arms: Gel Stent implantation
Procedure: Trabeculectomy — XEN Gel stent implantation either combined or as a stand-alone procedure
  Arms: Trabeculectomy

SUMMARY:
Trabeculectomy and XEN45 gel stent implantation are glaucoma surgeries that creates an aqueous humor (AH) shunt towards the subconjunctival space (filtration bleb). Once the AH reaches the subconjunctival space, it is removed by different paths such as the trans-bleb wall route. For this reason, the conjunctiva is considered an essential structure that may condition the glaucoma filtering procedures outcomes. As part of the inflammatory response, an unbalanced fibrosis during the postoperative period may lead to a bleb cavity scarring and failure; for this reason, bleb massage and antifibrotic injections (i.e., 5-Fluoruracil) are frequently required as part of the postoperative care of these procedures. There have been described several risk factors, such as intraocular pressure (IOP) lowering medications, previous surgical interventions or ocular surface disease that may predispose to an early failure. These preoperative factors fail to aim to predict the surgical outcomes.

However, ocular biomarkers may overcome this limitation. There are promising studies that have analyzed the role of in vivo confocal microscopy (IVCM), anterior-segment optical coherence tomography (AS-OCT) and conjunctival cytology impression as clinical tools that may improve the filtration bleb assessment at a cellular level.

DETAILED DESCRIPTION:
Detailed description Hypothesis

* Conjunctival biomarkers may represent a predictive factor to determine the XEN45 and trabeculectomy surgical success and outcomes
* A cellular-based analysis may help to predict postoperative pro-fibrotic changes that may lead to an early or mid-term surgery failure, and therefore it could help to improve the postoperative care of the filtering bleb.

Objective

* To evaluate the preoperative and postoperative conjunctival factors that may influence in the surgical outcomes of XEN45 gel stent compared to trabeculectomy using in vivo confocal microscopy, anterior segment optical coherence tomography and conjunctival cytology impression
* To assess the efficacy of XEN Gel stent and trabeculectomy to predict IOP, based on the morphologic characteristics of the filtering bleb
* To analyze the needling rate during the postoperative bleb management and the potential correlation to the pre and postoperative conjunctival changes and surgical success outcomes

Design Single-center, prospective, simple-blind study

Primary outcomes All the outcomes are measured pre and postoperative at each follow-up time

* In vivo confocal microscopy images: goblet cells density, dendritic cell density and stromal fibrosis
* Anterior segment optical coherence tomography: wall thickness and epithelium thickness
* Conjunctival cytology impression: dendritic cells, goblet cells

Secondary outcomes

* Intraocular pressure
* Number of IOP lowering medications
* Number of postoperative needling

Sample size calculation Based on the most assessed outcome in glaucoma surgeries and the only pilot study aiming to determine a similar outcome, to detect IOP differences between both procedures that may reflect the surgical outcomes of both procedures and therefore reflect the subconjunctival changes, accepting an alfa risk of 0.05 and a beta risk of 0.20 in a two-sided Student's T-test, 40 subjects are necessary in each group to recognize as statistically significant a difference greater than or equal to - 13,38 mm Hg in IOP, with a common standard deviation of 17%. A drop-out rate of 15% has been anticipated. If no drop-out rate is considered, the number of needed subjects is 68 (34 per group)

Method Single center, prospective, observational study of primary open angle glaucoma and uncontrolled intraocular pressure, progression of the disease confirmed by visual field examination that require either XEN gel stent implantation or trabeculectomy.

Preoperative examinations

* Medial records including ophthalmic procedures, other ocular diseases, intraocular pressure while on treatment, target pressure, visual field, detailed description of the optic disc, both preoperative and postoperative
* Glaucoma staging: peripapillary retinal nerve fiber layer, visual field (baseline, 3 moths and 6 months)
* Ocular biomarkers

  * In vivo confocal microscopy (baseline, 3 moths and 6 months)
  * Conjunctival impression cytology (baseline, 3 moths and 6 months)

A specific case report form (CRF) was designed with all variables and data required for the study, including potential complications

Surgery. Patients were assigned either to trabeculectomy or XEN stent implantation

Trabeculectomy: the surgical technique is as follows: retro/peribulbar o subtenon's anesthesia, superior corneal traction suture, phacoemulsification through 2.2 with in-the-bag IOL implantation, a fornix-based conjunctival flap, sufficient but not excessive cauterization, application mitomycin-C (MMC) 0,2 mg/ml for 2 minutes under the conjunctiva, then MMC was washed out with 100 ml of saline solution, then a scleral flap (4x3 mm in the trabeculectomy) is dissected. A sclerectomy with punch and peripheral iridectomy were performed, and suture nylon 10/00 sutures was used to place 3 or 4 stiches in the scleral flap

XEN gel stent: a clear cornea incision in the inferotemporal quadrant was performed, injecting the XEN 45 device into the superonasal quadrant using an ab interno approach. Approximately 15 min before inserting the implant, 0.1 ml of a MMC solution (0.01%) was injected into the superior conjunctiva. Both stand-alone and combined phaco-glaucoma procedures were used.

Post-operative treatment. All patients instilled ofloxacin antibiotic every 6 hours for 1 week, dexamethasone (every 2 hours for 1 month, every 4-6 hours on the second month and tapered during the third month according to surgeon's instructions). Atropine was also used when clinical finds recommended its use. Subconjunctival injections of anti-fibrotic agents (5-FU) and/or bleb needling were allowed and performed at the discretion of the surgeon

Statistical analysis

* Descriptive statistics, including mean and standard deviation for normally distributed variables and median and interquartile range for non-normally distributed variables, previous checked using Shapiro-Wilk test.
* Logistic regression models to evaluate the correlation with preoperative and postoperative factors and needling rate, surgical success (IOP < 18 mm Hg), and ocular biomarkers. The results will be reported as odds ratio (OR).
* All the reported values will be considered statistically significant at two-tailed p <0.05

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Written informed consent
* Older than 18 years old

Exclusion Criteria:

* Patients that don't fully understand the purpose and the postoperative care
* Severe or end-stage glaucoma
* Patients with prior ocular surgery, excluding uncomplicated phacoemulsification 6 months prior to the inclusion in the study

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
In vivo confocal microscopy of the filtering bleb | Preoperative to 6 months operative
  Increase of the mean microcysts density (MMD): number of cysts/mm2
Anterior segment optical coherence tomography microscopy of the filtering bleb | Preoperative to 6 months operative
  Differences in thickness of the conjunctival epithelial surface and the bleb wall, in micrometers
Conjunctival impression cytology of the filtering bleb | Preoperative to 6 months operative
  Increase in the percentage of goblet cells biomarkers

SECONDARY OUTCOMES:
Intraocular pressure | Preoperative to 6 months visit, at each follow-up visit
  Difference of intraocular pressure, in mm Hg
Glaucoma medications | Preoperative to 6 months visit, at each follow-up visit
  Difference between the number of glaucoma medications before and after each surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marta Pazos, MD, PhD, Principal Investigator — Hospital Clinic
Locations (1):
- Hospital Clínic - ICOF, Barcelona, Spain

REFERENCES:
- [Derived] Ventura-Abreu N, Molins B, Guerra-Meniconi J, Labay-Tejado S, Porto S, Muniesa MJ, Milla E, Pazos M. Longitudinal analysis of XEN45 gel stent bleb morphology using bleb grading scales, anterior segment-OCT, in vivo confocal microscopy, and impression cytology. Graefes Arch Clin Exp Ophthalmol. 2025 Oct 3. doi: 10.1007/s00417-025-06952-0. Online ahead of print. PMID 41042361